CLINICAL TRIAL: NCT06079034
Title: Impact of Cannulation Strategy on the Rate of Neurologic Injury in Infants With Respiratory Failure: A Propensity Score Analysis of the ELSO Registry
Brief Title: Impact of Cannulation Strategy on Neurologic Injury in Infants With Respiratory Failure
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Joseph Kohne (Pediatrics), Clinical Assistant Professor, University of Michigan
Other Study IDs: HUM00236110
Record Dates: First submitted 2023-09-22; First posted 2023-10-12 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Respiratory Failure
Keywords: ECMO
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Venovenous ECMO
  Interventions: Procedure: Venovenous ECMO
- Venoarterial ECMO
  Interventions: Procedure: Venoarterial ECMO

INTERVENTIONS:
Procedure: Venovenous ECMO — Initial support type of venovenous ECMO via a dual-lumen on two-site VV ECMO cannulation strategy
  Groups: Venovenous ECMO
Procedure: Venoarterial ECMO — Initial support type of venoarterial ECMO
  Groups: Venoarterial ECMO

SUMMARY:
There has been increasing use of venoarterial (VA) extracorporeal membrane oxygenation (ECMO) for infants with respiratory failure, up to 92% of neonatal respiratory support in 2021. This study seeks to leverage the increased use of VA ECMO in this cohort to enrich an evaluation of the differences in rate of intracranial hemorrhage and ischemic stroke between venovenous (VV) and VA ECMO among infants with respiratory failure where clinicians may choose either strategy.

This project is a retrospective review of data in the ELSO registry.

DETAILED DESCRIPTION:
From 2019-2021, there was increased use of venoarterial (VA) extracorporeal membrane oxygenation (ECMO) for infants with respiratory failure, up to 92% of neonatal respiratory support in 2021. The primary aim is to estimate the average effect on the rate of neurologic injury of VA ECMO versus venovenous (VV) among infants with respiratory failure over the period 2013-2018, during which clinicians could choose either cannulation strategy. This causal effect will be estimated using an inverse propensity weighted (IPW) approach. Secondarily, the investigators will project this estimated treatment effect forward into the period 2019-2021. The beginning of this period roughly corresponds to start of increased use of VA ECMO. Under the assumption of a homogenous treatment effect across both study periods, the rate of neurologic injury that would have occurred in 2019-2021 will be estimated, had the rate of VA ECMO not increased relative to pre-2019 levels. The hypothesis is that the results will point to an increased rate of neurologic injury starting in 2019 due to the increased use of VA ECMO.

ELIGIBILITY:
Inclusion Criteria:

* Patient weighed less than or equal to 10kg at start of ECMO
* Pulmonary support was the indication for ECLS
* Initial cannulation strategy was VV or VA
* The run occurred during the period 2013-2023

Exclusion Criteria:

* Patient had CDH
* Patient was post-cardiotomy
* Non-conventional initial cannulation strategies were employed, such as

  * Central Cannulation (surrogate for inability to achieve peripheral cannulation)
  * Veno-veno-arterial ECMO
  * Initial cannulation approach reported as "other"
* Patient was transported into or out of ELSO center on ECMO support
* Patient had pre-ECLS Cardiac Arrest
* Patient did not have subsequent ECMO runs in the ELSO registry

Min Age: 0 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients reported to the ELSO registry weighing less than or equal to 10 kilograms at the start of ECMO receiving ECMO for pulmonary support
Sampling Method: Non-Probability Sample
Enrollment: 5058 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Neurologic Injury | during critical illness supported by ECLS up to 14 days after ECLS stop time
  The outcome will be the composite occurrence of neurologic injury (ischemic stroke, intracranial hemorrhage, and brain death) that arises during critical illness supported by extracorporeal life support (ECLS) as reported to the Extracorporeal Life Support Organization (ELSO) registry, coded as a 0/1 variable (0 = no occurrence was reported during or after ECMO; 1 = one or more occurrence was reported).

SECONDARY OUTCOMES:
Mortality | through study completion (ECLS hospital discharge), an average of 2 months
  Whether a patient is discharged alive as reported to the ELSO registry
Duration of ECMO support | during the procedure (ECLS support)
  Hours of ECMO support as reported to the ELSO registry
Discharge Disposition | through study completion (ECLS hospital discharge), an average of 2 months
  Hospital discharge location as reported to the ELSO registry
Individual neurologic injury | during the procedure (ECLS support), and up to 14 days days after ECLS stop time
  For each neurologic injury included in the primary outcome measure, the injury will be assessed individually:
  proportion of patients with ischemic stroke as defined by the ELSO registry; proportion of patients with intracranial hemorrhage as defined by the ELSO registry; proportion of patients with brain death as defined by the ELSO registry

CONTACTS AND LOCATIONS:
Overall Officials: Joseph G Kohne, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Data received from the ELSO Registry is available to qualified researchers through an ELSO data request

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT06079034/SAP_000.pdf